CLINICAL TRIAL: NCT06895265
Title: Cross-Talk Between Arterial Calcifications
Brief Title: Potential Cross-Talk Between Arterial Calcifications
Acronym: PCTBAC
Status: Completed | Type: Observational
Sponsor: Ankara Ataturk Sanatorium Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Şahbender Koç, cardıologist, Ankara Ataturk Sanatorium Training and Research Hospital
Other Study IDs: 18.2.2024/66
Record Dates: First submitted 2025-02-26; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-02

CONDITIONS: Vascular Calcification; Atherosclerosis of Artery
Keywords: Vascular calcification
MeSH Terms: conditions — Vascular Calcification

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with abdominal CT records: The study group consisted of non-contrast abdominal CT records from 921 patients, aged between 40 and 90 years.

SUMMARY:
Potential Cross-Talk Between Arterial Calcifications Background Vascular calcification is a key component of atherosclerosis. This study investigates the potential correlations between aortic and coronary calcifications detected via abdominal CT, considering age-related variations, to explore the possibility of cross-talk.

Method A total of 921 patients (n=921) [male: 508 (55%), female: 413 (44.7%)] were divided into three age groups: 40-49, 50-69, and 70-90 years. Non-contrast abdominal CT scans were evaluated for calcifications in the coronary arteries, thoracic aorta, abdominal aorta (AA(1): suprarenal, AA(2): renal, AA(3): infrarenal), iliac arteries, and femoral artery. Aortic branches were categorized by calcification levels: none, <25%, 25-50%, ≥50%

DETAILED DESCRIPTION:
Atherosclerosis, a chronic inflammatory condition characterized by the buildup of plaque in the arteries, remains a major global health challenge. Vascular calcification (VC) is a critical component of atherosclerosis . VC can reduce the flexibility and compliance of the blood vessel wall, increase the instability of atherosclerotic plaque, and contribute to intravascular blood clotting, vascular obstruction, heart failure, and acute myocardial infarction. Furthermore, it can exacerbate cardiac workload .

Mediators from peripheral tissues, including inflammation and pro-inflammatory cytokines, are released into the circulation and may affect the heart. Coronary artery disease (CAD) also prompts the heart to release pro-inflammatory cytokines into the bloodstream. Cardiokines, which are heart-derived cytokines, can exert significant endocrine effects on other tissues, leading to damage in various peripheral organs .

Extracellular vesicles (EVs), which attach to receptor cell surfaces, can directly facilitate signal transmission or transfer their contents into the cell to elicit a functional response. EVs have been associated with subclinical atherosclerosis, which is diagnosed through ultrasound imaging of the femoral artery, carotid artery, or abdominal aorta . They have also been shown to play a role in the VC process. EVs facilitate communication between vascular wall cells and bone-vascular, liver-vascular, and adipose-vascular cells to regulate VC .

Understanding the relationship between calcification formations across different arterial regions is crucial for improving our knowledge of atherosclerosis pathophysiology and for facilitating the early diagnosis and follow-up of other affected regions. If such an association exists, it could provide valuable insights into systemic vascular diseases, ischemic patterns, and organ-specific perfusion dynamics.

Methods Patient selection and data collection Non-contrast abdominal CT records of 1,100 patients were reviewed. Records that included observable coronary sections starting from the aorta and femoral artery sections were included in the study. A total of 921 patients [male: 508 (55%), female: 413 (44.7%)] met the inclusion criteria and were divided into three age groups: 40-49, 50-69, and 70-90 years. Patients were classified into subgroups based on their medical records for Hypertension, Hyperlipidemia, Diabetes Mellitus, Coronary Artery Disease, and Chronic Obstructive Pulmonary Disease.

The CT records were retrospectively evaluated for calcifications in the coronary arteries, thoracic and abdominal aorta [AA] [suprarenal [1], renal [2], and infrarenal [3] segments], common iliac arteries [Communis], internal and external iliac arteries [Iliac], and femoral arteries.The CAC score is commonly used to quantify the extent of calcification across all coronary arteries and is typically categorized on a per-patient basis as None, Mild, Moderate, or Severe Following the examination of coronary lesions and the thoracic aorta for calcification, the abdominal aortic area was analyzed. Aortic calcifications were classified in horizontal cross-sectional slices, to some extent, in accordance with the classification proposed by Ehara et alRegional vessel segments were evaluated based on the extent of calcification and categorized as: none, <25%, 25-50%, and ≥50-100%.

ELIGIBILITY:
Inclusion Criteria:

Hypertension, Hyperlipidemia, Diabetes Mellitus, Coronary Artery Disease, Chronic Obstructive Pulmonary Disease

Exclusion Criteria:

Chronic renal failure Hemodialysis patients

-

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 40-90 with non-contrast abdominal CT records.
Sampling Method: Non-Probability Sample
Enrollment: 921 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Recording of coronary and abdominal aorta, as well as common, iliac, and femoral artery calcifications. | "Data were collected over a period of ten months."
  1-coronary artery calcifications, (CAC)] were visually classified in a simplified manner as either present or absent for a faster assessment 2-Following the examination of coronary lesions and the thoracic aorta for calcification, the abdominal aortic area was analyzed. Aortic calcifications were classified in horizontal cross-sectional slices.Regional vessel segments were evaluated based on the extent of calcification and categorized as: none, <25%, 25-50%, and ≥50-100%.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Atatürk Sanatoryum RTH, Ankara, Türki̇ye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared only upon reasonable request and approval by the study sponsor."
Supporting Information: SAP, CSR
Time Frame: De-identified individual participant data (IPD) and supporting information will be available starting 6 months after publication of study results. Data will be accessible for a period of 5 years.
Access Criteria: Researchers and qualified professionals will be able to access de-identified individual participant data (IPD) and supporting documents, including study protocols and statistical analysis plans. Data will be available through a secure online repository, requiring a formal data-sharing agreement and ethical approval
URL: ftp://sahbenderkoc@hotmail.com'